CLINICAL TRIAL: NCT02758054
Title: A Randomized Controlled Trial (RCT) of Patient Navigation for Lung Cancer Screening in an Urban Safety-Net System
Brief Title: Patient Navigation for Lung Cancer Screening in an Urban Safety-Net System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, David E Gerber, PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: STU 122015-046
Record Dates: First submitted 2016-04-25; First posted 2016-05-02 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Non-Small Cell Lung Carcinoma; Compliance Behavior; Prevention Harmful Effects
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Patient Compliance | interventions — Patient Navigation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants will experience standard practice for lung cancer early detection.
- Usual Care + Patient Navigation (Experimental): Participants will experience standard practice for lung cancer early detection plus the intervention.
  Interventions: Behavioral: Patient Navigation

INTERVENTIONS:
Behavioral: Patient Navigation — Patient navigated reminder calls containing information about screening appointments, reminders, hints to facilitate communication with physicians, and smoking cessation.
  Arms: Usual Care + Patient Navigation

SUMMARY:
The study proposes to evaluate a patient navigation intervention among a sample of 446 individuals referred for CT-based lung cancer screening in an urban safety-net setting.

DETAILED DESCRIPTION:
Widespread implementation of CT-based lung cancer screening is underway, but its impact on cancer morbidity and mortality can only be achieved IF people are screened at appropriate intervals and abnormal findings are appropriately assessed. The degree to which individuals, especially those from medically underserved populations with highest lung cancer risks, will adhere to the complex, multi-step process of CT-based lung cancer screening has emerged as a key question with immediate need for solution. Specific aims of the study are as follows:

* Aim 1: Compare rates of completion for clinically recommended steps in the lung cancer screening process between patients referred for CT-based lung cancer screening who are randomized to the navigation intervention versus patients who receive usual care.
* Aim 2: Compare changes in patient-reported outcomes, including satisfaction with care, psychosocial distress, and tobacco use between patients in the navigation intervention versus those who receive usual care for the CT-based lung cancer screening process.
* Aim 3 (Exploratory): Explore whether differences seen in Aims 1 and 2 are moderated theory-based patient attitudes and beliefs (perceived susceptibility, severity of lung cancer, perceived benefits/barriers to screening, self-efficacy).

This study will offer unprecedented insight into implementation of lung cancer screening for high-risk individuals in underserved settings. Findings will show whether navigation interventions increase adherence to the screening process and affect patient-reported outcomes among underserved populations. The proposed program aims to address these issues for lung cancer screening at its inception, rather than after disparities in screening uptake have already emerged.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for lung cancer screening using a low-dose CT scan modality who are considered high risk by USPSTF guidelines.
* Patients who speak English or Spanish

Exclusion Criteria:

* Patients who do not speak English or Spanish
* Patients who are or become ineligible as defined by USPSTF guidelines for lung cancer screening.

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Rate of Completion | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: David Gerber, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Lee SJC, Lee J, Zhu H, Chen PM, Wahid U, Hamann HA, Bhalla S, Cardenas RC, Natchimuthu VS, Johnson DH, Santini NO, Patel HR, Gerber DE. Assessing Barriers and Facilitators to Lung Cancer Screening: Initial Findings from a Patient Navigation Intervention. Popul Health Manag. 2023 Jun;26(3):177-184. doi: 10.1089/pop.2023.0053. Epub 2023 May 19. PMID 37219548
- [Derived] Gerber DE, Hamann HA, Santini NO, Abbara S, Chiu H, McGuire M, Quirk L, Zhu H, Lee SJC. Patient navigation for lung cancer screening in an urban safety-net system: Protocol for a pragmatic randomized clinical trial. Contemp Clin Trials. 2017 Sep;60:78-85. doi: 10.1016/j.cct.2017.07.003. Epub 2017 Jul 5. PMID 28689056